CLINICAL TRIAL: NCT04728152
Title: Evaluation of miRNAs in Endometriosis
Acronym: ENDOmiARN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Groupe expert en endometriose-6 centre expert en endometriose (Other)
Responsible Party: Principal Investigator, Sofiane Bendifallah, MD, PhD, Groupe expert en endometriose-6 centre expert en endometriose
Other Study IDs: n° Id-RCB 2020-A03297-32
Record Dates: First submitted 2021-01-23; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Endometriosis; Endometriosis Fertility; Endometriosis-related Pain
Keywords: endometriosis; miRNA
MeSH Terms: conditions — Endometriosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood and salivar test — Saliva samples will be taken (concomitant with a visit carried out as part of routine care):
  * At the pre-therapy visit (t3),
  * At the post-treatment visit (at 3-6 weeks).
  Blood samples will be taken at two stages (concomitant with a blood test performed as part of routine care):
  * At the pre-therapy visit (t3),
  * At the post-treatment visit (at 3-6 weeks).

SUMMARY:
We therefore propose a research project based on the prospective evaluation of miRNAs (blood and salivary) in patients with endometriosis diagnosed (by clinical examination and imaging) or suspected of endometriosis (clinical/radiological discordance) and in need of management in routine care (surgical or medical PMA) in the Endometriosis Expert Center Hospital.

ELIGIBILITY:
Inclusion Criteria:

- Patient aged 18 to 43 years old,

* Patient has dated and signed the consent form,
* Patient affiliated with the French health care system,
* Patients with formal endometriosis diagnosed by clinical examination and imaging or suspicion of endometriosis for which the diagnosis is a source of discrepancy between clinical and radiological data,
* Patient with an indication for medically assisted procreation (MAP) or surgery validated in CPR (in routine care),
* Patient who has had a pelvic MRI,
* Patient who completed the symptom and quality of life questionnaires

Exclusion Criteria:

* Pregnant patient,
* Patient infected with the human immunodeficiency virus (HIV),
* Patient with significant difficulties in reading or writing the French language,
* Patient with a personal history of cancer,
* Patient unable to comply with study and/or follow-up procedures,
* Patient who has objected to the collection of her data.
* Patient participating in another clinical research study.

Ages: 18 Years to 43 Years | Sex: Female
Age Groups: Adult
Study Population: The study population consists of women between the ages of 18 and 43 with a formal endometriosis diagnosis or suspicion of endometriosis.
  Patients in the study are already receiving routine medical (PMA) or surgical care in the Gynecology-Obstetrics and Reproductive Medicine Department of the hospital. All of these patients already benefit from a validation of therapeutic indications in a multidisciplinary consultation meeting (medical-surgical RCP or fertility).
  The patients concerned by the study are treated without any change in the course of care, nor modification of the therapeutic indications, nor modification of the diagnostic tests (imaging or biology) necessary according to the context, which are carried out according to the recommendations of the HAS.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-27 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Describe the evolution of miRNA expression (blood and salivary) | 1 month

SECONDARY OUTCOMES:
To quantify the reproducibility of salivary miRNA expression over time (between the inclusion visit and the pre-therapy visit) ; | 1 month
To describe (quantitatively and qualitatively) the expression of blood and salivary miRNAs in patients with suspected or actual endometriosis; | 1 time
Describe the expression of miRNAs (blood and salivary) according to the presence or absence of endometriosis and according to the endometriosis phenotype ; | 1 time
Describe the relationship between miRNA expression (blood and salivary) and the level of ovarian reserve, as estimated by the AMH assay in patients of childbearing age ; | 1 time

CONTACTS AND LOCATIONS:
Overall Officials: EMILE DARAI, PROF, Study Director — Centre Expert En Endométriose (C3E)
Locations (1):
- Sofiane Bendifallah, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dabi Y, Suisse S, Marie Y, Delbos L, Poilblanc M, Descamps P, Golfier F, Jornea L, Forlani S, Bouteiller D, Touboul C, Puchar A, Bendifallah S, Darai E. New class of RNA biomarker for endometriosis diagnosis: The potential of salivary piRNA expression. Eur J Obstet Gynecol Reprod Biol. 2023 Dec;291:88-95. doi: 10.1016/j.ejogrb.2023.10.015. Epub 2023 Oct 13. PMID 37857147